CLINICAL TRIAL: NCT05764083
Title: CSP #2028 - Epidemiology, Immunology and Clinical Characteristics of COVID-19 (EPIC3) Within the Veterans Health Administration
Brief Title: Epidemiology, Immunology and Clinical Characteristics of COVID-19 (EPIC3)
Acronym: EPIC3
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2028
Record Dates: First submitted 2023-03-08; First posted 2023-03-10 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: SARS-CoV-2; COVID-19
Keywords: Infectious disease; Chronic diseases; Critical care; Cohort; Epidemiologic; Observational; Prospective; Specimen banking; SARS-CoV-2; COVID-19
MeSH Terms: conditions — COVID-19; Communicable Diseases; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Biospecimen Retention: Samples With DNA — Nasopharyngeal swab, oropharyngeal swab, blood, saliva, stool, sputum, rectal swab, urine, and other residual clinical samples including cerebrospinal fluid and tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Inpatient Cohort: COVID-19-positive or -suspected inpatients: Eligible inpatient cohort participants include Veterans who receive inpatient care at VHA facilities and are tested for SARS-CoV-2. Members of this inpatient cohort include those with and without SARS-CoV-2 infection.
- Outpatient Cohort: COVID-19-positive or -suspected outpatients: Eligible outpatient cohort participants include Veterans who seek care in (1) VA medical center emergency departments, (2) VA medical center urgent care clinics, or (3) VA medical center COVID-19-specific testing sites, and who are tested for SARS-CoV-2 but do not require hospital admission at the time of evaluation. Members of this outpatient cohort include those with and without SARS-CoV-2 infection.
- Community Living Center Cohort: Community Living Center residents: Eligible Community Living Center cohort participants include all residents who reside in VA medical center-operated Community Living Centers. Members of this Community Living Center cohort include those with and without SARS-CoV-2 infection.

SUMMARY:
The purpose of this research is to gather information to answer questions about the Coronavirus Disease 2019 (COVID-19) which is caused by the Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection. This study will collect information and biological specimens from participants who have been tested for the SARS-CoV-2 infection. By doing this study, the investigators hope to learn important new information about SARS-CoV-2 infections and the potentially severe outcomes of COVID-19 to find better ways to manage and treat it in the future. The investigators also hope to learn what makes some people more susceptible to infection to help better inform Veterans on how to reduce their risk of infection. This study also involves the development and maintenance of a participant registry, a data repository, and a biorepository for future research.

DETAILED DESCRIPTION:
The objective of the study is to answer key research questions about the SARS-CoV-2 infection and COVID-19 natural history, clinical outcomes, and the development of immunity while also gathering biospecimens for future study as questions emerge about this new pathogen. The study is an observational cohort study of Veterans that is designed to gather longitudinal data on the epidemiology, virology, immunology, and clinical characteristics of the SARS-CoV-2 infection and COVID-19 disease during this early pandemic period while remaining flexible to the evolving needs of the Veterans Health Administration (VHA) system and emerging scientific questions. The study will enroll Veterans with and without SARS-CoV-2 infection in the inpatient, outpatient, and Community Living Center (CLC) extended care settings. Study procedures include questionnaires, clinical data abstraction from VHA electronic health records, and biological sampling. A key contribution of this study is to establish a research clinical and laboratory data repository and related research specimen repository, and participant registry for future studies of COVID-19, which is a newly emerging pandemic disease, and other health conditions. Finally, a long-term goal of this study is to provide the lessons learned from this COVID-19 pandemic to better anticipate and manage pandemics in the future for VHA and the general population.

There are 4 primary aims to this study: (1) identify patterns of SARS-CoV-2 viral shedding from multiple body sites in inpatient Veterans with COVID-19 infection during hospitalization through 28 days of follow-up; (2) characterize development of immunity among inpatient and outpatient Veterans with COVID-19 from the first VHA encounter through 24 months; (3) determine predictors of infection and disease course, severity and related death among inpatient and outpatient Veterans with and without SARS-CoV-2 infection and/or COVID-19 disease over 24 months; and (4) determine individual and health-facility-level risk factors for infection (including asymptomatic infection) with SARS-CoV-2 among Veterans at high risk for COVID-19 disease who are living in VHA Community Living Centers.

Veterans are likely to be substantially affected by COVID-19 due to a high prevalence of risk factors for severe COVID-19 disease. Understanding demographic, medical, and social factors that confer risk for severe COVID-19 disease is critical for improving care for Veterans with COVID-19. Characterizing viral shedding of SARS-CoV-2 infection during COVID-19 illness may yield important insight about factors that affect SARS-CoV-2 transmission. Characterizing the development of immunity among persons with COVID-19 is foundational to developing effective vaccines against the disease. Better understanding transmission risk and risk factors in the setting of VHA Community Living Centers will help prevent future infections.

ELIGIBILITY:
Inclusion Criteria:

* Eligible inpatient cohort participants include Veterans with confirmed, suspected, or unsuspected COVID-19 who receive inpatient care at VHA facilities
* Eligible outpatient cohort participants include Veterans who seek care in (1) VA medical center emergency departments, (2) VA medical center urgent care clinics, or (3) VA medical center COVID-19-specific testing sites, and who are tested for SARS-CoV-2 but do not require hospital admission at the time of evaluation
* Eligible Community Living Center cohort participants include all residents who reside in VA medical center-operated Community Living Centers

Exclusion Criteria:

* Veterans without a legally authorized representative who are unable to provide consent
* Potential participants who are not Veterans
* Veterans who are illiterate or have limited or no English language proficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is VA medical center inpatients, outpatients, and residents at Community Living Centers who meet the inclusion and exclusion criteria and are receiving healthcare at one of the VHA medical centers serving as study sites.
Sampling Method: Non-Probability Sample
Enrollment: 2824 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Health Status Change | Day 0 (enrollment) through 24 months
  Mortality

SECONDARY OUTCOMES:
Viral shedding | Day 0 (enrollment) through 6 months
  SARS-CoV-2 RNA from respiratory or gastrointestinal sampling sites
Immunity | Day 0 (enrollment) through 6 months
  SARS-CoV-2 IgM and IgG serum antibody titers

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Lee, MD PhD MA, Study Chair — VA Palo Alto Health Care System, Palo Alto, CA; Nicholas L. Smith, PhD, Study Chair — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected data may be shared dependent upon data safeguards and IRB approvals.
Supporting Information: ICF
Time Frame: Data will be made available for sharing 1 year after the publication of the last manuscript addressing the primary aims of the study.
Access Criteria: The VA Cooperative Studies Program (CSP) has a program for sharing CSP study data: Integrated Veteran Epidemiologic Study Data Resource (INVESTD-R). The INVESTD-R website is where information is provided on CSP studies with data that can be shared for secondary analyses or to support new data collection from study members who consented to be recontacted. Data will be shared with qualifying investigators at bona fide research institutions.
URL: https://www.vacsp.research.va.gov/CSPEC/Studies/INVESTD-R/CSP-2028-EPIC3.asp

REFERENCES:
- [Background] Huang L, Li X, Kamal SI, Sugimoto JD, Liu CH, Wang T, Morelli DK, Midthun JB, Pakanati VR, Deardorff KV, Sporleder JL, Lopez J, Holodniy M, Smith NL, Lee JS, Shah JA, Ross JM. Epidemiology, Immunology and Clinical Characteristics of COVID-19 (EPIC3)-Database of a prospective longitudinal observational study within the Veterans Health Administration. Front Public Health. 2025 Jun 2;13:1535315. doi: 10.3389/fpubh.2025.1535315. eCollection 2025. No abstract available. PMID 40538697
- [Result] Ross JM, Sugimoto JD, Timmons A, Adams J, Deardoff K, Korpak A, Liu C, Moore K, Wilson D, Bedimo R, Chang KM, Cho K, Crothers K, Garshick E, Gaziano JM, Holodniy M, Hunt CM, Isaacs SN, Le E, Jones BE, Shah JA, Smith NL, Lee JS; EPIC Investigators. Early Outcomes of SARS-CoV-2 Infection in a Multisite Prospective Cohort of Inpatient Veterans. Open Forum Infect Dis. 2023 Jun 27;10(7):ofad330. doi: 10.1093/ofid/ofad330. eCollection 2023 Jul. PMID 37484899
- [Result] Li X, Pakanati V, Liu C, Wang T, Morelli D, Korpak A, Baraff A, Isaacs SN, Vittor A, Chang KM, Le E, Smith NL, Lee JS, Ross JM, Shah JA; EPIC3 Investigators. Peripheral blood cytokine profiles predict the severity of SARS-CoV-2 infection: an EPIC3 study analysis. BMC Infect Dis. 2025 May 8;25(1):677. doi: 10.1186/s12879-025-10914-6. PMID 40340594
- See also: Seattle Epidemiologic Research and Information Center — http://www.seattle.eric.research.va.gov/
- See also: VA Cooperative Studies Program — http://www.research.va.gov/programs/csp/

DOCUMENTS (1):
  • Informed Consent Form (2021-11-26): https://cdn.clinicaltrials.gov/large-docs/83/NCT05764083/ICF_000.pdf